CLINICAL TRIAL: NCT02572050
Title: Assessment of a Robotic Distal Gastrectomy on Non-inferiority of N2 Area Nodal Dissection for Clinical Stage II or III Gastric Cancer
Brief Title: Assessment of a Robotic Distal Gastrectomy on Non-inferiority of N2 Area Nodal Dissection
Acronym: AaRon
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Keimyung University Dongsan Medical Center (Other); Seoul National University Hospital (Other); Seoul National University Bundang Hospital (Other); Samsung Medical Center (Other); Severance Hospital (Other); Ajou University School of Medicine (Other); Korea University (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, Young-Woo Kim, Professor, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2015-0191
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastroenterostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Robotic Distal Gastrectomy with D2 LND (Experimental): Robotic Distal Gastrectomy (RDG) with D2 LND for patient with stage II or III gastric cancer The primary efficacy endpoint of number of dissected lymph nodes in the N2 area (which is #7, #8a, #9, #11p and #12a according to the JRSSGC) after oncologic resection for clinical stage II or III gastric adenocarcinoma.assessment.
  Interventions: Procedure: Distal Gastrectomy with D2 LND

INTERVENTIONS:
Procedure: Distal Gastrectomy with D2 LND — Robotic Distal Gastrectomy with D2 lymphadenectomy(#7, #8a, #9, #11p, #12a in Japanese Classification) for patient with stage II or III gastric cancer
  Other Names: Robotic Distal Gastrectomy with D2 LND

SUMMARY:
Designed as a single arm multi-center prospective phase II trial, which evaluates the number of dissected lymph nodes in the N2-area as a surrogate parameter for adequate D2 lymphadenectomy in robotic distal gastrectomy (RDG) for clinical stage II or III gastric cancer.

DETAILED DESCRIPTION:
The number of retrieved LNs in the N2 area after RDG is going to be calculated according to the pathology reports and comparative analysis to a historic group undergone open surgery for clinical stage II or III gastric cancer at the NCC Korea last year.

METHODS AGAINST BIAS Minimizing selection bias: After initiation of the study, all patients will be screened consecutively and all eligible patients will be asked to enrol in the trial. The trial is designed as a prospective multi-center phase II trial. Patients are going to be allocated to RAG after giving signed consent after sufficient consideration time.

Minimizing performance bias: The study is planned as a prospective single arm multi-center trial, as the retrospective data suggest that there is no disadvantage in lymph node retrieval after RAG compared to LAG. Surgery is going to be performed according to the guidelines of the Japanese Research Society for the Study of Gastric Cancer (3rd edition). Japanese randomized controlled trials have proven effectiveness of adequate D2 lymphadenectomy in several randomized controlled trials. As number of dissected lymph nodes is a surrogate marker for adequate lymph node dissection, only patients with at least 25 lymph nodes removed (as obtained from pathology report) will be definitively included in the data assessment. Further lymph node stations No. #7, #8a, #9, #11p, #12a for subtotal gastrectomy according to the Japanese Guideline have to be dissected out of the surgical specimen and analyzed separately in the pathologic workup. All patients in the trial are going to be analyzed, as success rate of LN dissection in the N2-area is the primary endpoint. Surgery in the trial must be performed by a board certified surgeon who has taken part in a trial specific training course. Potential learning curve artefacts are negligible because the RAG is going to be performed by surgeons who are highly trained and experienced in robotic gastrectomy.

Participating surgeons should have experience as an operator of over 50 cases of open gastrectomy, over 50 laparoscopic gastrectomy, and over 15 cases of robotic gastrectomy. Furthermore, surgical quality will have to be enforced by intraoperative video documentation. Also, pictures of nodal dissection area after resection should be submitted to have a quality assurance.

Minimizing detection bias: Patients are going to regularly undergo standardized follow-up visits at 6, 12, 18, 24, 30, 36, 48, 60 months to be evaluated disease status with abdominopelvic CT. EGD will be done on 3, 12, 24, 36, 48 and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the stomach in patients that have not received any previous treatment for their cancer
* Tumours should be stage II or III according to the UICC 7th edition with no sign of distant metastasis and deemed resectable (R0) by the operating surgeon on preoperative staging by EGD, and CT of abdomen and pelvis
* Location of the tumor at the pylorus, antrum, angle, lower body and midbody to allow subtotal gastrectomy
* Age ≥ 19 years
* Written informed consent

Exclusion Criteria:

* Performance status ≥3
* Patients not eligible for surgery (ASA >=4)
* History of another primary cancer, except curatively treated in situ cervical cancer, curatively resected non-melanoma skin cancer. The inclusion of patients with other types of cancer that were successfully treated and did not recur within the last 5 years prior to study enrolment have to be discussed with the principal investigator.
* Evidence of distant metastasis on clinical staging
* Primary tumour deemed unresectable by operating surgeon
* Inadequate organ function as below

  * Bone marrow function defined as: (ANC ≤1.0x109/l, WBC (total) ≤ 2.5x109/l, Platelet Count ≤ 70x109/l, Haemoglobin ≤ 8 g/dl (can be post-transfusion)

    * Renal function with serum Creatinine ≥1.5 mg/dL) ③ Liver function defined as (Total Bilirubin≥ 2.0x (ULN), ALT/AST ≥2.5x ULN) ④ Coagulation profile: with PT (INR) ≥1.5, aPTT(sec) ≥1.5xULN
* Women of childbearing potential should have a negative pregnancy test within 7 days prior to commencing treatment, and must take adequate contraceptive precautions
* Simultaneous participation in another clinical trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of retrieved lymph nodes in the topographical N2 area | 1 week
  Number of retrieved lymph nodes in the topographical N2 area (#7, #8a, #9, #11p, #12a in Japanese Classification)

SECONDARY OUTCOMES:
Overall-survival | five years
  Overall-survival after five years of follow up
Recurrence-free survival | Three Year
  Three Year Recurrence-free survival
Incidence of local recurrence | Five Year
  Incidence of local recurrence
Early Complications | 1 month
  Early Complications( Abdominal wound complications , Fluid collection/intraabdominal abscess , Intraabdominal bleeding, Intraluminal bleeding, Anastomotic stenosis, Anastomotic leakage, Panceatic leakage, Pancreatitis, Atelectasis, Pneumonia, Urinary tract infection, Renal Dysfunction , Hepatic Dysfunction, Cardiac Disease ,Delayed gastric emptying : classified by Clavien-Dindo Classification(Definition and grading of complication) and be scored in accordance with the comprehensive complication index(http://assessurgery.com)
Late Complications | 5 year
  Late Complications(Intestinal Obstruction(Ileus), Anastomotic Stenosis, Iron Deficiency Anemia, etc.): classified by Clavien-Dindo Classification(Definition and grading of complication) and be scored in accordance with the comprehensive complication index(http://assessurgery.com)
Quality of life | 5 year
  Quality of life according to EQ-5

CONTACTS AND LOCATIONS:
Overall Officials: Young-Woo Kim, PhD, Principal Investigator — National Cancer Center of Korea
Locations (2):
- South Korea (2):
  - National Cancer Center of Korea, Goyang-si, Gyeonggi-do
  - Aju University Hospital, Suwon, Gyeonggi-do

REFERENCES:
- [Background] Cunningham D, Allum WH, Stenning SP, Thompson JN, Van de Velde CJ, Nicolson M, Scarffe JH, Lofts FJ, Falk SJ, Iveson TJ, Smith DB, Langley RE, Verma M, Weeden S, Chua YJ, MAGIC Trial Participants. Perioperative chemotherapy versus surgery alone for resectable gastroesophageal cancer. N Engl J Med. 2006 Jul 6;355(1):11-20. doi: 10.1056/NEJMoa055531. PMID 16822992
- [Result] Song J, Oh SJ, Kang WH, Hyung WJ, Choi SH, Noh SH. Robot-assisted gastrectomy with lymph node dissection for gastric cancer: lessons learned from an initial 100 consecutive procedures. Ann Surg. 2009 Jun;249(6):927-32. doi: 10.1097/01.sla.0000351688.64999.73. PMID 19474671
- [Result] Woo Y, Hyung WJ, Pak KH, Inaba K, Obama K, Choi SH, Noh SH. Robotic gastrectomy as an oncologically sound alternative to laparoscopic resections for the treatment of early-stage gastric cancers. Arch Surg. 2011 Sep;146(9):1086-92. doi: 10.1001/archsurg.2011.114. Epub 2011 May 16. PMID 21576595
- [Result] Eom BW, Yoon HM, Ryu KW, Lee JH, Cho SJ, Lee JY, Kim CG, Choi IJ, Lee JS, Kook MC, Rhee JY, Park SR, Kim YW. Comparison of surgical performance and short-term clinical outcomes between laparoscopic and robotic surgery in distal gastric cancer. Eur J Surg Oncol. 2012 Jan;38(1):57-63. doi: 10.1016/j.ejso.2011.09.006. Epub 2011 Sep 25. PMID 21945625
- [Result] Yoon HM, Kim YW, Lee JH, Ryu KW, Eom BW, Park JY, Choi IJ, Kim CG, Lee JY, Cho SJ, Rho JY. Robot-assisted total gastrectomy is comparable with laparoscopically assisted total gastrectomy for early gastric cancer. Surg Endosc. 2012 May;26(5):1377-81. doi: 10.1007/s00464-011-2043-0. Epub 2011 Nov 16. PMID 22083338
- [Result] Kitano S, Shiraishi N, Uyama I, Sugihara K, Tanigawa N; Japanese Laparoscopic Surgery Study Group. A multicenter study on oncologic outcome of laparoscopic gastrectomy for early cancer in Japan. Ann Surg. 2007 Jan;245(1):68-72. doi: 10.1097/01.sla.0000225364.03133.f8. PMID 17197967
- [Result] Huscher CG, Mingoli A, Sgarzini G, Sansonetti A, Di Paola M, Recher A, Ponzano C. Laparoscopic versus open subtotal gastrectomy for distal gastric cancer: five-year results of a randomized prospective trial. Ann Surg. 2005 Feb;241(2):232-7. doi: 10.1097/01.sla.0000151892.35922.f2. PMID 15650632
- [Result] Noshiro H, Shimizu S, Nagai E, Ohuchida K, Tanaka M. Laparoscopy-assisted distal gastrectomy for early gastric cancer: is it beneficial for patients of heavier weight? Ann Surg. 2003 Nov;238(5):680-5. doi: 10.1097/01.sla.0000094302.51616.2a. PMID 14578729
- [Result] Kim YW, Baik YH, Yun YH, Nam BH, Kim DH, Choi IJ, Bae JM. Improved quality of life outcomes after laparoscopy-assisted distal gastrectomy for early gastric cancer: results of a prospective randomized clinical trial. Ann Surg. 2008 Nov;248(5):721-7. doi: 10.1097/SLA.0b013e318185e62e. PMID 18948798
- [Result] Uyama I, Kanaya S, Ishida Y, Inaba K, Suda K, Satoh S. Novel integrated robotic approach for suprapancreatic D2 nodal dissection for treating gastric cancer: technique and initial experience. World J Surg. 2012 Feb;36(2):331-7. doi: 10.1007/s00268-011-1352-8. PMID 22131088
- [Result] Sasako M, Sano T, Yamamoto S, Kurokawa Y, Nashimoto A, Kurita A, Hiratsuka M, Tsujinaka T, Kinoshita T, Arai K, Yamamura Y, Okajima K; Japan Clinical Oncology Group. D2 lymphadenectomy alone or with para-aortic nodal dissection for gastric cancer. N Engl J Med. 2008 Jul 31;359(5):453-62. doi: 10.1056/NEJMoa0707035. PMID 18669424
- [Result] Sakuramoto S, Sasako M, Yamaguchi T, Kinoshita T, Fujii M, Nashimoto A, Furukawa H, Nakajima T, Ohashi Y, Imamura H, Higashino M, Yamamura Y, Kurita A, Arai K; ACTS-GC Group. Adjuvant chemotherapy for gastric cancer with S-1, an oral fluoropyrimidine. N Engl J Med. 2007 Nov 1;357(18):1810-20. doi: 10.1056/NEJMoa072252. PMID 17978289
- [Result] Lakatos E, Lan KK. A comparison of sample size methods for the logrank statistic. Stat Med. 1992 Jan 30;11(2):179-91. doi: 10.1002/sim.4780110205. PMID 1579757
- [Result] Com-Nougue C, Rodary C, Patte C. How to establish equivalence when data are censored: a randomized trial of treatments for B non-Hodgkin lymphoma. Stat Med. 1993 Jul 30;12(14):1353-64. doi: 10.1002/sim.4780121407. PMID 8210831
- See also: The official web site of National Cancer Center — http://www.ncc.re.kr